CLINICAL TRIAL: NCT05057104
Title: Non-inferiority Study of Unresectable Hepatocelluar Carcinoma Receiving Stereotactic Radiotherapy Combined With Hepatic Arterial Chemoembolization Compared With Conversion Hepatectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SBRTplusTACE VS. HR
Record Dates: First submitted 2021-09-13; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Hepatocellular Carcinoma Non-resectable; Conversion
Keywords: CyberKnife; unresectable hepatocelluar carcinoma; TACE; hepatectomy; prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CK-SBRT with TACE group
- Conversion hepatectomy after CK-SBRT plus TACE

SUMMARY:
To compare the prognosis and adverse reactions of unresectable hepatocellular carcinoma receiving stereotactic radiotherapy combined with hepatic arterial chemoembolization and conversion hepatectomy

ELIGIBILITY:
Inclusion Criteria:

* Unresectable HCC patients were diagnosed by a surgeon and/or radiologist and oncologist according to the international guidelines for the management of HCC or by pathology
* Patients who received SBRT plus TACE have tumor regression, and surgical experts assess that R0 resection could be achieved
* CP-A or B classification;
* Eastern Cooperative Oncology Group (ECOG) score 0-1;
* Platelet count≥50 × 109/L, white blood count≥1.5 × 109/L;
* ICG R15≤10%;
* Normal effective liver volume >30%;
* patients infected with hepatitis B virus who are treated with adefovir or entecavir; patients infected with hepatitis C virus whose HCV DNA are negative.

Exclusion Criteria:

-the patients receive other treatments (such as targeted treatment, immune checkpoint inhibitors,etc) after CK-SBRT plus TACE.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unresectable HCC patients meet surgical criteria after CK-SBRT plus TACE.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2021-10-10 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival time | From date of randomization until the date of death from any cause, assessed up to 24 months.

SECONDARY OUTCOMES:
Progression-free survival time | From date of randomization until the date of disease progression or date of death from any cause, whichever came first, assessed up to 24 months.
Radiation-induced liver injury rates | From the date of radiotherapy completion until the 4 months after therapy,up to 6 months.
Adverse reaction | From the date of radiotherapy completion until the 4 months after therapy,up to 6 months

REFERENCES:
- [Background] Erratum: Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2020 Jul;70(4):313. doi: 10.3322/caac.21609. Epub 2020 Apr 6. No abstract available. PMID 32767693
- [Background] Su TS, Lu HZ, Cheng T, Zhou Y, Huang Y, Gao YC, Tang MY, Jiang HY, Lian ZP, Hou EC, Liang P. Long-term survival analysis in combined transarterial embolization and stereotactic body radiation therapy versus stereotactic body radiation monotherapy for unresectable hepatocellular carcinoma >5 cm. BMC Cancer. 2016 Nov 3;16(1):834. doi: 10.1186/s12885-016-2894-9. PMID 27809890
- [Background] Wei X, Jiang Y, Zhang X, Feng S, Zhou B, Ye X, Xing H, Xu Y, Shi J, Guo W, Zhou D, Zhang H, Sun H, Huang C, Lu C, Zheng Y, Meng Y, Huang B, Cong W, Lau WY, Cheng S. Neoadjuvant Three-Dimensional Conformal Radiotherapy for Resectable Hepatocellular Carcinoma With Portal Vein Tumor Thrombus: A Randomized, Open-Label, Multicenter Controlled Study. J Clin Oncol. 2019 Aug 20;37(24):2141-2151. doi: 10.1200/JCO.18.02184. Epub 2019 Jul 8. PMID 31283409
- [Background] Rim CH, Kim CY, Yang DS, Yoon WS. Comparison of radiation therapy modalities for hepatocellular carcinoma with portal vein thrombosis: A meta-analysis and systematic review. Radiother Oncol. 2018 Oct;129(1):112-122. doi: 10.1016/j.radonc.2017.11.013. Epub 2017 Dec 9. PMID 29233562
- [Background] Lau WY, Ho SK, Yu SC, Lai EC, Liew CT, Leung TW. Salvage surgery following downstaging of unresectable hepatocellular carcinoma. Ann Surg. 2004 Aug;240(2):299-305. doi: 10.1097/01.sla.0000133123.11932.19. PMID 15273555
- [Background] Tomonari T, Sato Y, Tanaka H, Tanaka T, Taniguchi T, Sogabe M, Okamoto K, Miyamoto H, Muguruma N, Saito Y, Imura S, Bando Y, Shimada M, Takayama T. Conversion therapy for unresectable hepatocellular carcinoma after lenvatinib: Three case reports. Medicine (Baltimore). 2020 Oct 16;99(42):e22782. doi: 10.1097/MD.0000000000022782. PMID 33080748
- [Background] Hoffe SE, Finkelstein SE, Russell MS, Shridhar R. Nonsurgical options for hepatocellular carcinoma: evolving role of external beam radiotherapy. Cancer Control. 2010 Apr;17(2):100-10. doi: 10.1177/107327481001700205. PMID 20404793
- [Background] Chiang CL, Chan ACY, Chiu KWH, Kong FS. Combined Stereotactic Body Radiotherapy and Checkpoint Inhibition in Unresectable Hepatocellular Carcinoma: A Potential Synergistic Treatment Strategy. Front Oncol. 2019 Nov 12;9:1157. doi: 10.3389/fonc.2019.01157. eCollection 2019. PMID 31799176